CLINICAL TRIAL: NCT06424847
Title: Effects of a Lifestyle and Sleep Intervention Program on Quality of Life and Physical Activity Levels in Non-exercising Adults, SPIRAL+ Randomized Controlled Trial
Brief Title: Effects of a Lifestyle and Sleep Intervention in Non-exercising Adults
Acronym: SPIRAL+
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPIRAL+
Record Dates: First submitted 2024-04-25; First posted 2024-05-22 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Inactivity, Physical; Lifestyle Risk Reduction
Keywords: lifestyle intervention; sleep intervention; physical activity; behavior change techniques
MeSH Terms: conditions — Sedentary Behavior; Risk Reduction Behavior; Motor Activity | interventions — Exercise; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lifestyle intervention (physical activity and diet) (Active Comparator)
  Interventions: Behavioral: Lifestyle intervention (physical activity and diet)
- Lifestyle (physical activity and diet) and Sleep intervention (Active Comparator)
  Interventions: Behavioral: Lifestyle (physical activity and diet) and Sleep intervention
- Health education intervention (Sham Comparator)
  Interventions: Behavioral: Health education intervention

INTERVENTIONS:
Behavioral: Lifestyle intervention (physical activity and diet) — The physical activity intervention will be based on validated behavior change theories aimed at the initiation and long-term maintenance of physical activity.
  Participants will be referred to specialists in Adapted Physical Activity for a 6-month program. Exercise sessions will include aerobic exercise and muscle strengthening exercises. Participants will participate in one supervised sessions per week. They will receive instructions for exercising on their own on the other days in order to reach physical activity guidelines. They will also receive instructions and tips to limit sedentary behavior and increase their physical activity throughout the day.
  Participants will benefit from an initial consultation with a dietitian and 4 follow-up visits. The follow-up visits will be either group-based or individual, based on participants choice and availabilities. Dietary recommendations will be based on public health guidelines in France aimed at eating a healthy, balanced diet.
  Arms: Lifestyle intervention (physical activity and diet)
Behavioral: Lifestyle (physical activity and diet) and Sleep intervention — Participants will benefit from the physical activity and diet intervention detailed above and the following sleep intervention. Participants will fill out an online sleep diagnostic tool includes validated sleep questionnaires (Pittsburgh Sleep Quality Index, Epworth sleepiness scale, Insomnia Severity Index, Berlin questionnaire, Horne and Ostberg questionnaire).
  Participants will also log their sleep habits in a 14-day sleep diary. Based on the sleep specialists' review of the results of the questionnaires, sleep diary and analysis of sleep-wake patterns, participants who require further exploration will be referred to a sleep specialist for a consultation and if necessary the appropriate treatment for their sleep disorder.
  All participants in this group will benefit from an individualized sleep hygiene intervention. They will benefit from a baseline interview and 3 follow-up visits.
  Arms: Lifestyle (physical activity and diet) and Sleep intervention
Behavioral: Health education intervention — Participants randomized to the control group will benefit from a health education intervention in order to limit deception bias.
  Arms: Health education intervention

SUMMARY:
Background. Cardiovascular diseases (CVDs) are the leading cause of premature mortality and disability accounting for one third of all deaths worldwide with considerable impacts on economics and on quality of life. Recent studies suggest that a lifestyle intervention might have a role in the reduction of CDV risk. Lifestyle intervention programs typically combine physical activity, diet and behavior modification components. Poor sleep health is highly prevalent in the general population and contributes to increased risk of several noncommunicable diseases. However, sleep is rarely addressed in lifestyle intervention programs in primary prevention. Given the high prevalence of poor sleep health in people without a diagnosed sleep disorder, and the associated health consequences, there is a clear need for broad-reaching, effective interventions to improve sleep quality in subclinical populations.

Aims. The main objective of this study is to compare a lifestyle intervention program including a sleep intervention compared to a lifestyle intervention program alone on the health-related quality of life (measured by the EQ-5D-5L) and physical activity levels of non-exercising adults.

Methods. Non-exercising adults (n=201) will be recruited in the community via advertisement or their primary care doctor and then randomized to one of the following 3 groups : lifestyle intervention, lifestyle and sleep intervention or standard care. The lifestyle intervention includes a physical activity component (physical activity initiation visit and 6 months of supervised physical activity, once weekly), a diet component (consultation with a dietician and 3 group sessions). The sleep intervention includes individualized face-to-face sessions aimed at improving and optimizing sleep hygiene.

At baseline and after 6 and 12 months, quality of life, physical activity levels, cardiovascular and metabolic risk factors will be evaluated.

Perspectives. This study should determine whether adding a sleep intervention dimension to a lifestyle intervention program provides significant benefits in terms of quality of life and physical activity levels. Based on this study, the modalities of real-life lifestyle intervention programs could be reconsidered in order to provide optimal primary prevention.

ELIGIBILITY:
Inclusion Criteria:

* Participant who is physically inactive (i.e. less than 150 minutes of moderate intensity physical activity per week)
* Participant aged 18 to 80 years old
* Participant able to provide written informed consent
* Participant able to participate in regular physical activity (no medical contraindication to exercise)
* Participant affiliated to social security or a similar regimen

Exclusion Criteria:

* Any condition that in the opinion of the responsible physician or investigator makes the potential participant unsuitable for the study
* A participant who scores 11111 on the EQ-5D-5L questionnaire
* A diagnosed and treated sleep disturbance (sleep apnea, insomnia, restless legs syndrome)
* Persons concerned by articles L1121-5, L1121-6 and L1121-8 of the public health code (i.e. pregnancy, person deprived of liberty or subject to a legal protection measure, vulnerable person or legally protected adult)
* Person already included in another interventional study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Steps per day | 6 months after randomization
  Measured using an activity monitor (Actigraph)
Health-related quality of life | 6 months after randomization
  EuroQol (Europe Quality of Life) EQ-5D-5L questionnaire.The EQ-5D-5L is a brief, multiattribute, generic, health status measure composed of 5 questions with Likert response options (descriptive system). The descriptive system covers 5 dimensions of health (mobility, self-care, usual activities, pain or discomfort, and anxiety or depression) with 5 levels of severity in each dimension (no problems, slight problems, moderate problems, severe problems, and unable to perform or extreme problems). The worst health state is (55555) and the best health state is (11111).

SECONDARY OUTCOMES:
Subjective sleep quality | Baseline, 6 months and 12 months
  Pittsburg Sleep Quality Index. The Pittsburgh Sleep Quality Index (PSQI) contains 19 self-rated questions and 5 questions rated by the bed partner or roommate (if one is available). Only self-rated questions are included in the scoring. The 19 self-rated items are combined to form seven "component" scores, each of which has a range of 0-3 points. In all cases, a score of "0" indicates no difficulty, while a score of "3" indicates severe difficulty. The seven component scores are then added to yield one "global" score, with a range of 0-21 points, "0" indicating no difficulty and "21" indicating severe difficulties in all areas.
Sleep duration | Baseline, 6 months and 12 months
  Measured using an activity monitor (Actigraph GT3X) and Sunrise sleep
Sleep quality | Baseline, 6 months and 12 months
  Measured using an activity monitor (Actigraph GT3X) and Sunrise
Modrate to vigorous intensity physical activity time | Baseline, 6 months and 12 months
  Time spent in moderate-to-vigorous physical activity measured by a physical activity monitor, Actigraph GT3X
Light intensity physical activity time | Baseline, 6 months and 12 months
  Time spent in light intensity physical activity measured by a physical activity monitor, Actigraph GT3X
Vigorous intensity physical activity time | Baseline, 6 months and 12 months
  Time spent in vigorous intensity physical activity measured by a physical activity monitor, Actigraph GT3X
Sedentary time | Baseline, 6 months and 12 months
  Sedentary time measured by a physical activity monitor Actigraph GT3X
Cardiorespiratory fitness (VO2peak) | Baseline, 6 months and 12 months
  Cardiorespiratory stress test
6 minute walk test distance | Baseline, 6 months and 12 months
  Six-minute walk test: This test measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes (the 6MWD)
24-hr systolic and diastolic blood pressure | Baseline, 6 months and 12 months
  Measured using an ambulatory BP device
Health-related quality of life | Baseline, 6 months and 12 months
  EuroQol (Europe Quality of Life) EQ-5D-5L questionnaire.The EQ-5D-5L is a brief, multiattribute, generic, health status measure composed of 5 questions with Likert response options (descriptive system). The descriptive system covers 5 dimensions of health (mobility, self-care, usual activities, pain or discomfort, and anxiety or depression) with 5 levels of severity in each dimension (no problems, slight problems, moderate problems, severe problems, and unable to perform or extreme problems). The worst health state is (55555) and the best health state is (11111).
Body composition | Baseline, 6 months and 12 months
  Measured using bio-electrical impedance
Grip strength | Baseline, 6 months and 12 months
  Measured using a dynamometer
Quality of life SF-36 | Baseline, 6 months and 12 months
  The 36-Item Short Form Health Survey questionnaire measures eight scales: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH). The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Anxiety symptoms | Baseline, 6 months and 12 months
  General Anxiety Disorder-7 (GAD-7) questionnaire. The score is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." GAD-7 total score for the seven items ranges from 0 to 21.
Depressive symptoms | Baseline, 6 months and 12 months
  Patient Health Questionnaire-9 (PHQ-9). Each item is evaluated on a severity scale ranging from 0 to 3 where the respondent is asked to rate how often each symptom occurred over the last 2 weeks (0-not at all; 1-several days; 2-more than half of the days or 3-nearly every day), yielding a total score ranging from 0-27.
Mental well-being | Baseline, 6 months and 12 months
  Warwick-Edinburgh Mental Wellbeing Scale. The Likert scale represents a score for each item from 1 to 5 respectively, giving a minimum score of 14 and maximum score of 70. All items are scored positively. The overall score for the WEMWBS is calculated by totalling the scores for each item, with equal weights.
Motivation toward physical activity | Baseline, 6 months and 12 months
  Motivation Scale towards Health-Oriented Physical Activity questionnaire. A higher score indicates higher motivation towards physical activity.
Social deprivation | Baseline, 6 months and 12 months
  Social deprivation score. This questionnaire is designed to assess the level of precariousness by the means of 11 binary items. Among these 11 items, two are very frequent in material deprivation scales: items #4-5. Six are related to social deprivation: items #1, #3, #6-9. One is related to health and financial difficulties: item #1. The last two [#10-11] are specific to precariousness scales. The final score can vary from 0 (no precariousness), to 100 (extreme precariousness), each item having its own weight.
Eating behavior | Baseline, 6 months and 12 months
  The Dutch Eating Behavior Questionnaire (DEBQ) is a 33-item self-report questionnaire that is aimed to assess three distinct eating behaviors in adults: (1) emotional eating, (2) external eating, and (3) restrained eating. Items on the DEBQ range from 1 (never) to 5 (very often), with higher scores indicating greater endorsement of the eating behavior.
Insomnia Severity | Baseline, 6 months and 12 months
  Insomnia Severity Index. The total score is the sum of all seven items. Total score ranges from 0-28. A higher score indicates more symptoms of insomnia.
Subjective sleepiness | Baseline, 6 months and 12 months
  Epworth Sleepiness Score. The ESS is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. Most people engage in those activities at least occasionally, although not necessarily every day. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life (ASP), or their 'daytime sleepiness'.
Attitude towards physical activity practice | Baseline, 6 months and 12 months
  This scale measures the main psychological predictors of physical activity according to the theory of planned behaviour. Attitude is measured by 5 items. A higher score indicates more a favorable attitude.
Self-efficacy | Baseline, 6 months and 12 months
  This scale measures the main psychological predictors of physical activity according to the theory of planned behaviour. Self-efficacy is measured by 3 items, a higher score indicates higher self-efficacy.
Subjective norms | Baseline, 6 months and 12 months
  This scale measures the main psychological predictors of physical activity according to the theory of planned behaviour. Subjective norms is measured by 2 items, a higher score indicates more favorable subjective norms.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Coudurier, MD, Principal Investigator — MCoudurier3@chu-grenoble.fr
Locations (1):
- Grenoble University Hospital, Grenoble, France